CLINICAL TRIAL: NCT06803615
Title: The Use of Beat-to-Beat Noninvasive 3D Mapping to Study Patients Candidates for Concomitant Surgical Ablation for Persistent and Long-standing Persistent Atrial Fibrillation
Brief Title: Noninvasive Mapping Before Surgical Ablation
Acronym: NIMSA
Status: Active, not recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Emilio Osorio, MD, Principal Investigator, Medical University of Vienna
Other Study IDs: 1046/2018
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Atrial Fibrillation; Electrocardiographic Imaging; Noninvasive Mapping; Surgical Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Electrocardiographic imaging — Electrocardiographic imaging is an electrophysiological mapping technique which is used to noninvasively map cardiac arrhythmias.
  Other Names: Noninvasive surface mapping; Noninvasive mapping; Beat-to-beat noninvasive 3D mapping

SUMMARY:
The purpose of this study is to assess the electrophysiological mechanism of atrial fibrillation by means of a beat-to-beat noninvasive 3D mapping method in patients with concomitant persistent and long-standing persistent atrial fibrillation undergoing surgical ablation.

ELIGIBILITY:
Inclusion Criteria:

* legal age (18-90a)
* life expectancy > 2 years
* patients suffering from persistent and long standing atrial fibrillation
* scheduled for concomitant surgical ablation
* possibility to follow-up
* given informed consent

Exclusion Criteria:

* vulnerable patient groups
* pregnancy
* any previous surgical ablation
* acute surgical indications
* any physical condition that leads to a life expectancy of less than two years
* any contraindication to the treatments necessary for the trial's conduction as e.g.

  * known allergic reaction to contrast agent
  * known allergic reaction to antiarrhythmic drugs
  * claustrophobia or anxiety in small spaces
  * severe renal impairment
  * unmanageable hyperthyroidism
* participation in any other clinical trial that either excludes enrolment or may be a confounding factor to results
* voluntary retention

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with persistent or long-standing persistent atrial fibrillation scheduled for concomitant surgical ablation at Vienna General Hospital of the Medical University of Vienna.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
The patients electrophysiological mapping results acquired with ECGI will be analyzed: Number and distribution of rotor and focal activities will be measured. | Prior to the planned procedure.
  The primary objective of this study is to measure the patients electrophysiological mapping results acquired with ECGI, namely the number and distribution of focal and rotor activities.

OTHER OUTCOMES:
Freedom from AF during 12 and 24 months of follow-up. | From surgery until 24 months after the procedure.
  A pre-specified outcome measure is to measure freedom from AF during 12 and 24 months of follow-up. The impact of the preoperative mapping results and the applied respective ablation technique will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Osorio, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared on reasonable request to the principal investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From 03/2025 until 12/2025

REFERENCES:
- [Derived] Osorio-Jaramillo E, Conci L, Schloglhofer T, Coti I, Strassl A, Schukro C, Zimpfer D, Ehrlich MP, Ad N. Electrocardiographic Imaging as Preoperative Tool in Persistent and Long-Standing Persistent Atrial Fibrillation: A Prospective Observational Study. Interdiscip Cardiovasc Thorac Surg. 2025 Sep 1;40(9):ivaf198. doi: 10.1093/icvts/ivaf198. PMID 40828886